CLINICAL TRIAL: NCT05603598
Title: LEAP2 on Postprandial Glucose Metabolism and Food Intake in Obese Males
Brief Title: LEAP2 on Postprandial Glucose Metabolism and Food Intake n Obese Males
Acronym: LEAP2-OBCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, MD, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-19038628
Record Dates: First submitted 2022-10-19; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — liver-expressed antimicrobial peptide 2, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): IV infusion of saline, approximately 5.5 hours
  Interventions: Drug: LEAP-2 Protein, Human
- Liver-enriched antimicrobial peptide 2 (Experimental): IV infusion of LEAP2, approximately 5.5 hours
  Interventions: Drug: LEAP-2 Protein, Human

INTERVENTIONS:
Drug: LEAP-2 Protein, Human — Intravenous infusion, mixed meal test, ad libitum meal test

SUMMARY:
The study aims to delineate the effects of the naturally occurring peptide liver-enriched antimicrobial peptide 2 (LEAP-2) on postprandial glucose metabolism and food intake in obese volunteers. The overall objective is to investigate the physiological importance of LEAP-2 in obese subjects.

DETAILED DESCRIPTION:
In a recent study, the molecular phenotype of enteroendocrine cells in the small intestine before and after Roux-en-Y Gastric Bypass (RYGB) surgery in obese individuals was examined. Enteroendocrine cells were identified and isolated from intestinal biopsies and analysed for differentially expressed genes by Illumina High Throughput RNA-sequencing. It was discovered that the gene encoding liver-enriched antimicrobial peptide 2 (LEAP-2), a naturally occurring peptide in humans, was significantly upregulated compared to baseline expression. Interestingly, LEAP-2 was recently shown to antagonize ghrelin function in response to feeding in mice. Moreover, the mature murine LEAP-2 peptide is identical in mice and humans. Thus, LEAP-2 has been identified as an endogenous peptide that may be able to alter feeding behaviour and maintenance of glucose levels during calorie restriction. Our group recently found a 12 % relative reduction in ad libitum food intake and reduced postprandial glucose excursions.

The present study hypothesis is that LEAP-2 alters postprandial glucose metabolism and decreases appetite as well as food intake in relation to a liquid mixed meal and a standardised ad libitum meal compared with saline (placebo) in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men
* Age between 18 and 25 years
* Body mass index between 30-50 kg/m2
* Informed consent

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary and/or gastrointestinal disorder(s)
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Allergy or intolerance to ingredients included in the standardised meals
* First-degree relatives with diabetes and/or glycated haemoglobin (HbA1c) >48 mmol/mol
* Regular tobacco smoking or use of other nicotine-containing products
* Any ongoing medication that the investigator evaluates would interfere with trial participation.
* Any physical or psychological condition that the investigator evaluates would interfere with trial participation including any acute or chronic illnesses

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on self-representation
Enrollment: 20 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Food intake, kilojoules | 290 to 320 minutes
  Difference in food intake during an ad libitum meal. Food intake is examined as kilojoules of food eaten during the ad libitum meal.
Food intake, kilojoules per kilogram body weight | 290 to 320 minutes
  Difference in food intake during an ad libitum meal. Food intake is examined as kilojoules per kilogram body weight of food eaten during the ad libitum meal.

SECONDARY OUTCOMES:
VAS, appetite | -35 to 320 minutes
  Visual analogue scales (VASs) assessing appetite (from 0 to 9,5 cm on a scale = from minimum to maximum sensation)
VAS, satiety | -35 to 320 minutes
  Visual analogue scales (VASs) assessing satiety sensations (from 0 to 9,5 cm on a scale = from minimum to maximum sensation)
VAS, hunger | -35 to 320 minutes
  Visual analogue scales (VASs) assessing hunger sensations (from 0 to 9,5 cm on a scale = from minimum to maximum sensation)
VAS, thirst | -35 to 320 minutes
  Visual analogue scales (VASs) assessing thirst (from 0 to 9,5 cm on a scale = from minimum to maximum sensation)
Alterations in gastric emptying | -35 to 320 minutes
  Paracetamol concentration in plasma after intake of 1.5 g paracetamol
Plasma insulin levels and beta cell secretion assessed by plasma C-peptide concentration relative to plasma glucose concentration | -35 to 320 minutes
  Plasma insulin levels and beta cell secretion assessed by plasma C-peptide concentration relative to plasma glucose concentration
Plasma/serum concentrations of LEAP-2, acyl-ghrelin as well as other glucose- and appetite-regulating gut hormones | -35 to 320 minutes
  Plasma/serum concentrations of LEAP-2, acyl-ghrelin as well as other glucose- and appetite-regulating gut hormones
Changes in resting energy expenditure (REE) | -35 to 320 minutes
  Changes in resting energy expenditure (REE) measured by indirect calorimetry
Triglyceride responses | -35 to 320 minutes
  Plasma triglyceride
Cholesterol responses | -35 to 320 minutes
  Plasma Cholesterol
Free fatty acid responses | -35 to 320 minutes
  Plasma Free fatty acid

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Capital Region, Denmark